CLINICAL TRIAL: NCT06094608
Title: IBD-Sleep: A Pilot Study Looking at Changes in Sleep Timing and IBD Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Helen Burgess, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00234262; 1R01DK136520 (NIH)
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to study arm. The PI, study coordinator and research assistants will remain unblinded to perform safety assessments and provide feedback on intervention adherence. Blinded staff will wear buttons as an upfront visual cue to remind participants not to talk about their treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Morning light treatment (Experimental): A 1 hour per day morning light treatment starting at average wake time, or up to 1 hour earlier to accommodate the morning schedule. The daily treatment continues for 4 weeks.
  Interventions: Device: Morning light treatment
- Treatment-as-usual (Active Comparator): Participants will be instructed to continue to follow their usual sleep schedule for 4 weeks.
  Interventions: Behavioral: Treatment-as-usual

INTERVENTIONS:
Device: Morning light treatment — Light therapy via the Re-Timer. Participants will conduct light treatment in the mornings at home for one hour using Re-timer®.
  Other Names: Re-Timer®
  Arms: Morning light treatment
Behavioral: Treatment-as-usual — Participants will not make modifications to their activities or sleep schedule.
  Arms: Treatment-as-usual

SUMMARY:
This research study is testing whether changes in sleep timing and morning light treatment may have an impact on symptoms related to inflammatory bowel disease.

DETAILED DESCRIPTION:
This study will test a consumer health light therapy device (Re-Timer) for people with inflammatory bowel disease to better understand how it affects IBD-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven IBD
* Active IBD symptoms
* Impaired IBD quality of life
* Age >/=18 years old
* Fluency in English
* Physically able to travel for study visits

Exclusion Criteria:

* Ileostomy, colostomy, ileoanal pouch, or ileorectal anastomoses, are planned for imminent surgery and/or have short bowel syndrome
* Other significant chronic disease
* Retinal pathology, history of eye surgery, taking photosensitizing medications
* Recent history of light treatment
* Lifetime psychotic or bipolar disorder
* Acute suicidal ideation
* Substance use disorder in the past 3 months, cannabis use >1/week
* High risk for or diagnosed with obstructive sleep apnea, and/or narcolepsy
* Severe hearing problem, intellectual disability or serious cognitive impairment
* Pregnant, trying to get pregnant, or breastfeeding
* Night work or travel outside the eastern time zone in the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Short IBD Questionnaire (SIBDQ) score | Baseline, post-treatment approximately 36 days
  SIBDQ is 10 questions, each with a Likert like scale with 7 options and lower scores indicate poorer quality of life.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire 9 (PHQ-9) score | Baseline, post-treatment approximately 36 days
  PHQ-9 is a depression score ranging from 0 through 27. No depression 0-4, mild 5-9, moderate 10-14, moderately severe 15-19, severe 20-27.
Change in Patient-Reported Outcomes Measurement Information System Sleep Disturbance (PROMIS) Short-Form 8b | Baseline, post-treatment approximately 36 days
  PROMIS Sleep Disturbance measures self-reported sleep quality during the past seven days. The measure includes 8-items with higher scores indicating greater sleep disturbance.
For patients with Crohn's Disease (CD) - Change in Harvey Bradshaw Index (HBI) | Baseline, post-treatment approximately 36 days
  The HBI is a clinician-rated measure of disease severity in Crohn's disease (CD). The HBI has items addressing a range of symptoms including general well-being, abdominal pain, liquidity/softness of stool, presence of an abdominal mass and complications. The total score reflects the following: score <5 = remission, 5 to 7 = mild disease activity, 8 to 16 = moderate disease activity and >16 = severe disease activity.
For patients with Ulcerative Colitis (UC) - Change in Simple Clinical Colitis Activity Index (SCCAI) | Baseline, post-treatment approximately 36 days
  The SCCAI is a clinician-rated measure of disease severity in ulcerative colitis (UC). The SCCAI has items addressing a range of symptoms from bowel frequency, defecation urgency, blood in stool, general well-being, and other extracolonic disease features. Scores range from 0 to 19 points, and scores < or equal to 2.5 indicate clinical remission.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Burgess, Ph.D., Principal Investigator — University of Michigan; Cathy Goldstein, M.D., M.S., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are open to sharing data by any appropriate mechanism indicated by NIH program staff.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After scientific papers are accepted for publication and the data will be available for 7 years after study completion.
Access Criteria: Researchers requesting data will first have to sign a data sharing agreement, agreeing to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, electronically securing the data while in use, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, no use of the data for commercial purposes and proper acknowledgement of the data resource.

REFERENCES:
- [Derived] Cohen-Mekelburg S, Goldstein CA, Rizvydeen M, Fayyaz Z, Patel PJ, Berinstein JA, Bishu S, Cushing-Damm KC, Kim HM, Burgess HJ. Morning light treatment for inflammatory bowel disease: a clinical trial. BMC Gastroenterol. 2024 May 22;24(1):179. doi: 10.1186/s12876-024-03263-2. PMID 38778264